CLINICAL TRIAL: NCT03082300
Title: A Phase 1, Randomized, 2-period Crossover Study to Assess Bioequivalence of a Tablet Formulation Versus a Capsule Formulation of ASP8273 in Subjects With Non-small Cell Lung Cancer Harboring Epidermal Growth Factor Receptor Mutations
Brief Title: A Study of ASP8273 in Subjects With Non-small Cell Lung Cancer (NSCLC) Harboring Epidermal Growth Factor Receptor (EGFR) Mutations
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Following recommendation by SOLAR Study IDMC, Astellas closed enrollment in ASP8273 studies.
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 8273-CL-0112
Record Dates: First submitted 2017-03-13; First posted 2017-03-17 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Non-small Cell Lung Cancer (NSCLC); Epidermal Growth Factor Receptor (EGFR) Mutations
Keywords: ASP8273; Epidermal growth factor receptor (EGFR) mutations; naquotinib; Non-small cell lung cancer (NSCLC); Bioequivalence
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — naquotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Pharmacokinetic phase: ASP8273 Tablet then Capsule Sequence (Experimental): Subjects will receive a single oral dose in tablet formulation on Day 1 of period 1 under fasted condition, then subjects will receive a single oral dose of ASP8273 in capsule formulation on Day 1 of period 2 under fasted condition. Each period will be for 5 days
  Interventions: Drug: naquotinib
- Pharmacokinetic phase: ASP8273 Capsule then Tablet Sequence (Experimental): Subjects will receive a single oral dose in capsule formulation on Day 1 of period 1 under fasted condition, then subjects will receive a single oral dose of ASP8273 in tablet formulation on Day 1 of period 2 under fasted condition. Each period will be for 5 days
  Interventions: Drug: naquotinib
- Postpharmacokinetic phase: ASP8273 Capsule Formulation (Experimental): All subjects will receive ASP8273 capsules in once-daily dosing for 1 cycle (28 days)
  Interventions: Drug: naquotinib

INTERVENTIONS:
Drug: naquotinib — Oral
  Other Names: ASP8273

SUMMARY:
The objective of this study is to evaluate the bioequivalence of a tablet formulation versus a capsule formulation of ASP8273 following a single dose under fasted condition in subjects with non-small cell lung cancer (NSCLC) harboring epidermal growth factor receptor (EGFR) mutations. The study will also evaluate the safety and tolerability of a tablet formulation as a single dose and a capsule formulation as a single and multiple dose of ASP8273 in subjects with NSCLC harboring EGFR mutations.

DETAILED DESCRIPTION:
Study and subjects will be divided into two phases: a pharmacokinetic (PK) and a postpharmacokinetic phase. The pharmacokinetic phase will follow a randomized, 2 period, 2 sequence single dose crossover design. Each period will be 5 days in duration. Within the sequence, both an ASP8273 tablet and ASP8273 capsule will be administered under fasted condition. The postpharmacokinetic phase will consist of up to 1 cycle (28 days) of continuous once daily dosing in post PK phase with ASP8273 capsules. Dose modifications are allowed if necessary in post PK phase and they follow a step-wise dose reduction. Subject is able to re-escalate dose level if reaction is stable.

ELIGIBILITY:
Inclusion Criteria:

* Subject has histologically confirmed locally advanced or unresectable Stage IIIB (not amenable to receive curative treatments such as chemo-radiation)/IV or metastatic NSCLC.
* Subject has Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.
* Subject has an EGFR activating mutation based on local testing.
* Subject has predicted life expectancy ≥ 12 weeks.
* Subject must meet all of the following criteria on the laboratory tests. In case of multiple laboratory data within this period, the most recent data should be used.

  * Neutrophil count > 1000/mm^3
  * Platelet count ≥ 7.5 x 10^4/mm^3
  * Hemoglobin > 8.0 g/dL
  * Serum creatinine <2.0 x upper limit of normal (ULN) or estimated glomerular filtration rate of > 50 mL/min as calculated by the Cockcroft Gault Method
  * Total bilirubin < 1.5 × ULN (except for subjects with documented Gilbert's syndrome)
  * AST (Aspartate aminotransferase (GOT) and ALT (Alanine aminotransferase (GPT)) < 3.0 × ULN (upper limit of normal) or ≤ 5 × ULN if subject has documented liver metastases
  * Serum sodium level ≥ 130 mmol/L
* Subject agrees not to participate in another interventional study while receiving study drug and participating in the present study.
* Female subject must either:

  * Be of nonchildbearing potential:
  * Postmenopausal (defined as at least 1 year without any menses) prior to screening, or
  * Documented surgically sterile (e.g., hysterectomy, bilateral salpingectomy, bilateral oophorectomy) Or, if of childbearing potential,
  * Agree not to try to become pregnant during the study and for 28 days after the final study drug administration
  * And have a negative blood pregnancy test at the time of screening
  * And if heterosexually active, agrees to consistently use 1 form of highly effective birth control* starting at screening and throughout the study period and for 28 days after the final study drug administration.
* Female subject must agree not to breastfeed at screening and throughout the study period, and for 28 days after the final study drug administration.
* Female subject must not donate ova starting at screening and throughout the study period, and for 28 days after the final study drug administration.
* A sexually active male subject with female partner(s) who are of childbearing potential is eligible if:

  * Agrees to use a male condom starting at screening and continue throughout study treatment and for 90 days after the final study drug administration. If the male subject has not had a vasectomy or is not sterile as defined below their female partner(s) is utilizing 1 form of highly effective birth control*starting at screening and continue throughout study treatment and for 90 days after the male subject receives their final study drug administration.
* Male subject with a pregnant or breastfeeding partner(s) must agree to remain abstinent or use a condom for the duration of the pregnancy or time partner is breastfeeding throughout the study period and for 90 days after the final study drug administration
* Male subject must not donate sperm starting at screening and throughout the study period, and for 90 days after the final study drug administration.
* Subject must be willing to fast for approximately 10 hours predose and 4 hours postdose on day 1 of each period in the pharmacokinetic phase.

  * Highly effective forms of birth control include:

    * Consistent and correct usage of established hormonal contraceptives that inhibit ovulation,
    * Established intrauterine device or intrauterine system.
    * Vasectomy (A vasectomy is a highly effective contraception method provided the absence of sperm has been confirmed. If not, an additional highly effective method of contraception should be used).
    * Male subject is sterile due to a bilateral orchiectomy.

Exclusion Criteria:

* Subject has an ongoing toxicity ≥ Grade 2 (NCI CTCAE Version 4.03) attributable to prior medication to treat solid tumor (except alopecia) at screening.
* Subject has received investigational therapy within 28 days or 5 half-lives, whichever is longer, prior to the first dose of study drug.
* Subject has received treatment with any other agent with antitumor activity including chemotherapy, radiotherapy, or immunotherapy within 14 days as well as EGFR tyrosine kinase inhibitor within 6 days prior to first dose of study drug.
* Subject has any of the following within 14 days prior to the first dose of study drug:

  * Major surgical procedure (other than study related biopsy), or a major surgical procedure is planned to occur during the planned study duration
  * Blood transfusions or hemopoietic factor therapy
  * Evidence of active infection requiring systemic therapy
* Subject has symptomatic central nervous system (CNS) metastasis. Subject with previously treated brain or CNS metastases is eligible provided that the subject has recovered from any acute effects of radiotherapy and is not requiring systemic steroids and any whole brain radiation therapy was completed at least 2 weeks prior to study drug administration, or any stereotactic radiosurgery was completed at least 1 week prior to study drug administration.
* Subject has a known history of a positive test for human immunodeficiency infection.
* Subject has a known history of a positive test for hepatitis B surface antigen or hepatitis C antibody.
* Subject has known history of serious hypersensitivity reaction to ASP8273, or any component of the formulation used.
* Subject has severe or uncontrolled systemic diseases including uncontrolled hypertension or active bleeding diatheses.
* Subject has history of drug-induced interstitial lung disease (ILD) or any evidence of active ILD.
* Subject has ongoing cardiac arrhythmia that is Grade ≥ 2 or uncontrolled atrial fibrillation of any grade.
* Subject currently has Class III or IV New York Heart Association congestive heart failure.
* Subject has history of severe/unstable angina, myocardial infarction or cerebrovascular accident within 6 months prior to the planned first dose of study drug.
* Subject has active gastrointestinal ulcer or gastrointestinal bleeding within 3 months prior to the planned first dose of study drug.
* Subject has concurrent corneal disorder or any ophthalmologic condition that makes the subject unsuitable for study participation (e.g., advanced cataracts, glaucoma).
* Subject has difficulty taking oral medication or any digestive tract dysfunction or inflammatory bowel disease that would interfere with the intestinal absorption of drug.
* Subject has another past or active malignancy that requires treatment. Prior carcinoma in situ and/or nonmelanoma skin cancer after curative resection are permitted.
* Subject has received the following within 14 days prior to the first dose of study drug:

  * Strong or moderate CYP3A4 inhibitors or inducers
  * Strong or moderate P-gp inhibitors or inducers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2017-03-24 (Actual); Primary Completion 2017-05-12 (Actual); Study Completion 2017-06-19 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of ASP8273 in plasma: Cmax | Up to Day 5 in each period of Phase 1 (maximum of 10 days)
  Cmax: Maximum plasma concentration. Pharmacokinetic phase only
Pharmacokinetics of ASP8273 in plasma: AUCinf | Up to Day 5 in each period of Phase 1 (maximum of 10 days)
  AUCinf: Area under the concentration time curve extrapolated to time infinity. Pharmacokinetic phase only
Pharmacokinetics of ASP8273 in plasma: AUClast | Up to Day 5 in each period of Phase 1 (maximum of 10 days)
  AUClast: Area under the concentration time curve from time zero to the last quantifiable concentration. Pharmacokinetic phase only
Pharmacokinetics of ASP8273 in plasma: AUC72 | Up to Day 5 in each period of Phase 1 (maximum of 10 days)
  AUC72: Area under the concentration time curve truncated at 72 hours. Pharmacokinetic phase only

SECONDARY OUTCOMES:
Pharmacokinetics of ASP8273 in plasma: t1/2 | Up to Day 5 in each period of Phase 1 (maximum of 10 days)
  t1/2: Terminal elimination half-life. Pharmacokinetic phase only
Pharmacokinetics of ASP8273 in plasma: tmax | Up to Day 5 in each period of Phase 1 (maximum of 10 days)
  tmax: The time of maximum concentration. Pharmacokinetic phase only
Pharmacokinetics of ASP8273 in plasma: tlast | Up to Day 5 in each period of Phase 1 (maximum of 10 days)
  tlast: The time of last observed concentration. Pharmacokinetic phase only
Pharmacokinetics of ASP8273 in plasma: CL/F | Up to Day 5 in each period of Phase 1 (maximum of 10 days)
  CL/F: Oral clearance. Pharmacokinetic phase only
Pharmacokinetics of ASP8273 in plasma: Vz/F | Up to Day 5 in each period of Phase 1 (maximum of 10 days)
  Vz/F: Apparent volume of distribution. Pharmacokinetic phase only
Safety and tolerability assessed by nature, frequency, and severity of adverse events (AES) | Up to day 30
  For both pharmacokinetic and postpharmacokinetic phases
Number of participants with vital sign abnormalities and/or adverse events related to treatment | Up to day 30
  Vital signs include systolic and blood diastolic pressure, temperature and pulse rate. For both pharmacokinetic and postpharmacokinetic phases
Number of participants with laboratory abnormalities and/or adverse events related to treatment | Up to day 30
  Laboratory values include biochemical, hematological, coagulation and urine analysis. For both pharmacokinetic and postpharmacokinetic phases
Safety assessed by routine 12-lead electrocardiograms (ECG) | Up to day 30
  Routine 12-lead ECGs will be performed after the subject has been in a supine position for at least 5 minutes. For both pharmacokinetic and postpharmacokinetic phases

CONTACTS AND LOCATIONS:
Overall Officials: Senior Medical, Study Director — Astellas Pharma Global Development, Inc.
Locations (3):
- United States (3):
  - Beverly Hills Cancer Center, Beverly Hills, California
  - Renovatio Clinical, The Woodlands, Texas
  - US Oncology - Virginia Cancer Specialists, P.C. (VCS), Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- See also: Link to results on the Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/study.aspx?ID=251